CLINICAL TRIAL: NCT05332483
Title: The Effect of Megestrol Acetate on Grade 2 Endometrioid Endometrial Cancer in Patients Waiting for Definitive Surgery, a Prospective Trial
Brief Title: Study of Megestrol Acetate in Grade 2 Endometrioid Endometrial Cancer
Acronym: MA-EEC
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Ontario Institute for Cancer Research (Other)
Responsible Party: Principal Investigator, Bojana Djordjevic, Staff gynecologic pathologist, Sunnybrook Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4858
Record Dates: First submitted 2022-04-10; First posted 2022-04-18 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-11

CONDITIONS: Endometrial Cancer
Keywords: Endometrial endometrioid carcinomas; Oral progestin therapy; Fertility sparing treatment; Predictive biomarkers
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Megestrol Acetate; Megestrol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arm 1 - Megestrol (Experimental): All study participants will receive Megestrol acetate, 160 mg daily (two 40mg tablets twice a day), for a minimum of 18 days.
  Interventions: Drug: Megestrol Acetate

INTERVENTIONS:
Drug: Megestrol Acetate — Megestrol acetate, 160 mg daily (two 40mg tablets twice a day), for a minimum of 18 days.
  Other Names: MEGESTROL; Megace

SUMMARY:
This is a single centre, single arm, open label, preoperative window of opportunity study. Grade 2 endometrioid endometrial carcinoma patients awaiting surgery will be prospectively recruited to receive a pre-operative progestin therapy course. Therapy response will be histologically evaluated and correlated with clinical and molecular data by comparison of responders vs. non-responders pre- and post-treatment tumor samples.

DETAILED DESCRIPTION:
The incidence of endometrial cancer is increasing due to the rising rates of obesity. Further, the average age at onset is decreasing. As a result, there is a growing interest in fertility-sparing treatments, such as progesterone-based therapy. While the role of progestins for the conservative management of atypical hyperplasia and with Fédération Internationale de Gynécologie et d'Obstétrique (FIGO) grade 1 endometrial endometrioid carcinomas (EEC), assigned on preoperative endometrial biopsy, is well established, there is limited clinical experience in patients FIGO grade 2 EECs (EEC2) for whom the current standard therapy is hysterectomy. However, there are case reports of successful progestin treatment of patients with preoperative biopsy EEC2, suggesting that progestin response mechanisms are functional in select EEC2s and that hormonal treatment may be a viable option if the responsive patients could be safely identified.

In this study, the investigators will prospectively recruit EEC2 patients for pre-operative progestin treatment. Participants will be given high-dose progestin from day of consent for a minimum of 21 days. This will allow investigators to generate a unique cohort of matched pre-progestin treatment biopsies and post-treatment surgical specimens for each participant. The investigators intend to analyze clinical, pathological and transcriptomic data of EEC2 that histologically respond to progestin therapy versus their counterparts that do not, with the goal of identifying candidate predictive biomarkers and clinical parameters that would supplement pathological screening of these lesions to better stratify patient classification to good and poor responders. Once good responders are successfully characterize, this will enable the investigators to identify patients with biopsy EEC2 that could be safely managed conservatively with oral progestin therapy. For young patients, who have not completed their family planning, this could mean the difference between undergoing a hysterectomy versus retaining their fertility.

ELIGIBILITY:
Inclusion Criteria:

* Adult female patient 18 years of age or older.
* Confirmed diagnosis of FIGO grade 2 endometrioid endometrial cancer on preoperative endometrial biopsy read by a pathologist with a subspecialty in gynecologic pathology.
* Stage 1 endometrioid endometrial cancer on preoperative endometrial biopsy.
* P53 wild type immunohistochemistry on preoperative endometrial biopsy.
* Patients eligible for primary staging surgery for definitive treatment for their cancer.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Required Initial Laboratory Values obtained within 3 days of enrolment following standard of care protocols: Absolute Neutrophil Count (ANC) ≥ 1,500/mm3; Platelet Count ≥ 100,000/mm3; eGFR ≥ 60 mL/min/1.73m2; Total Bilirubin ≤ 1.5 x upper limit of normal (ULN); AST / ALT ≤ 2.5 x upper limit of normal (ULN).
* Informed consent for this study is obtained and signed by the participant or have an acceptable Substitute Decision Maker (SDM) capable of signing the informed consent form on behalf of the participant.

Exclusion Criteria:

* Patients cannot be receiving systemic or hormonal therapy for treatment of the endometrial cancer.
* Prior radiation therapy for treatment of the endometrial cancer is not allowed.
* Stage 2 or 3 endometrioid endometrial cancer on preoperative endometrial biopsy.
* Abnormal p53 immunohistochemistry on preoperative endometrial biopsy.
* History of an allergic reaction to medroxyprogesterone acetate.
* History of venous thromboembolic event (including previous deep vein thrombosis or pulmonary embolism).
* Family history of venous thromboembolic event.
* Have a >20 pack-year smoking history.
* Patients unwilling or unable to follow the study protocol schedule.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-07-05 (Actual); Primary Completion 2023-10-12 (Actual); Study Completion 2023-10-12 (Actual)

PRIMARY OUTCOMES:
Overall response rate of patients with biopsy grade 2 endometrioid endometrial cancer treated preoperatively with Megestrol acetate for a minimum of 21 days. | 2 years
  Tumor response will be strictly histologically defined. Surgical specimens of each patient will be grossed in the pathology department as per standard of care.
  The degree of tumor response will be defined as follows:
  * Complete response: resolution of both cytologic atypia and architectural complexity to resemble non-tumorous endometrium.
  * Partial response: resolution of cytologic atypia and/or decrease in tumor grade (ie. From FIGO grade 2 to FIGO grade 1)
  * No response: persistence of the original lesion or progression to higher tumor grade.

SECONDARY OUTCOMES:
Correlations between response to progestin and clinical, histological and transcriptomic pre-operative biomarkers that may impact therapy planning. | 3 years
  The secondary outcome answers whether there is a pre-treatment biomarker signature at baseline biopsy that can predict therapeutic response to progestin among grade 2 endometrioid endometrial cancer patients. To identify molecular correlates of treatment response transcriptional profiling of pre-treatment and post-treatment tissue specimens will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Bojana Djordjevic, MD, Principal Investigator — Sunnybrook Health Sciences Centre; Danielle Vicus, MD, MSc, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences, Toronto, Ontario, Canada